CLINICAL TRIAL: NCT02794402
Title: A Parallel, Double-blinded, Randomized, 6 Months, Two Arms Study With Lifestyle Intervention and Bydureon® or Lifestyle Intervention and Placebo in Adolescents With Obesity to Explore Differences With Regard to Change in BMI SDS
Brief Title: Double-blinded, 6 Months Study With Bydureon® or Placebo in Adolescents With Obesity to Explore Changes in BMI
Acronym: Combat-JUDO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Peter Bergsten, Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-001628-45
Record Dates: First submitted 2016-05-17; First posted 2016-06-09 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bydureon (Active Comparator): s.c. once Weekly
  Interventions: Drug: Exenatide
- Placebo (Placebo Comparator): s.c. once Weekly
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Drug: Exenatide — Bydureon (Exenatide once weekly) injections s.c.
  Arms: Bydureon
Behavioral: Placebo — Placebo once weekly injections sc
  Arms: Placebo

SUMMARY:
Combat-JUDO (Combating Juvenile Diabetes and Obesity through normalization of beta-cell function) is part of a collaborative project funded by the Seventh Framework Programme of the European Commission aiming to develop innovative therapeutic strategies by increasing pharmacology-based alternatives targeting insulin hypersecretion for the treatment of young obese individuals.

The prevalence of childhood obesity is ranging between 5-25% in Europe. The reason behind these alarming figures is mostly a changing environment with a more sedative lifestyle and supply of excess food. However, specific gene mutations have also been linked to obesity and new genes are continuously being discovered. There are very few effective means of intervention in children with obesity available today. Obesity is closely associated with a number of related metabolic diseases and some children with obesity develop the metabolic syndrome at an early stage in life. Individuals with obesity have an increased risk of developing type 2 diabetes mellitus (T2DM) and with the current increase in childhood obesity, some children will develop T2DM already in their adolescent years with huge impact on their long-term health and life expectancy.

Lifestyle modification interventions, including behavioural treatment, diet modification and physical activity, are cornerstones of primary and secondary prevention/treatment of pediatric obesity today. Exenatide is a GLP-1 (glucagon-like peptide-1) receptor agonist approved for use in adults with T2DM to improve glycemic control. A pilot study with exenatide treatment in non-diabetic children and adolescents with severe obesity showed a reduced BMI of approximately 5% and improved markers of insulin resistance and β-cell function were observed.

The Combat-JUDO study is a parallel, double-blind, randomized study comparing lifestyle intervention + exenatide 2 mg vs lifestyle and intervention + placebo in adolescents with obesity. The lifestyle intervention includes regular nutritional and psychological support at 4 occasions during the study as well as physical activity on a weekly basis. Exenatide/placebo is given as a subcutaneous injection once weekly for 24 weeks. The primary objective of the study is to compare the change in BMI-SDS (according to WHO) from baseline to the 6 months visit between the two treatment arms.

The study includes males and females of age 10-18 years and 5 months with BMI SDS >2.0 or age-adapted BMI >30 kg/m2.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-specific procedures.
2. Males or females of age 10-18 years and 5 months.
3. Obesity (BMI SDS > 2.0 or age-adapted BMI > 30 kg/m2), according to WHO.
4. Not sexually active or usage of adequate anticonception. Female subjects must also have negative pregnancy tests. Methods that can achieve a failure rate of less than 1% per year (Pearl index <1), when used consistently and correctly, are considered as highly effective birth control methods. Such methods include:

   * Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

     * oral
     * intravaginal
     * transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation:

     * oral
     * injectable
     * implantable
   * Intrauterine device (IUD)
   * Intrauterine hormone-releasing system (IUS)
   * Bilateral tubal occlusion
   * Vasectomised partner Sexual abstinence (if refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the preferred and usual lifestyle of the subject). 5. Ability to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Known syndromal obesity, such as Prader-Willi syndrome, Laurence-Moon syndrome or Bardet-Biedl syndrome.
2. Pregnancy or lactation.
3. Indigestion-causing diseases.
4. Severe gastrointestinal disease.
5. Total or partial gastric or small intestine resection.
6. Type 1 or Type 2 diabetes mellitus.
7. Kidney disease (acute or chronic, according to physician (Creatinin/Urea/Cystatin-C for Schwartz Calculation)).
8. Hypo-/Hyperthyroidism, unless under stable treatment.
9. Severe Vitamin D insufficiency, unless under stable treatment.
10. Abnormal QT interval.
11. Clinically significant abnormal laboratory values, e.g. Triglycerides > 400 mg/dl (Salzburg) or > 4,5 mmol/L (Uppsala), Amylase > 300 U/L (Salzburg) or > 5,1 µkat/L (Uppsala), Lipase > 180 U/L (Salzburg) or > 15 µkat/L (Uppsala) or Calcitonin > 11.7 pg/ml (Salzburg) or > 3,4 pmol/L (Uppsala) for females and > 17 pg/ml (Salzburg) or > 5,0 pmol/L (Uppsala) for males.
12. Severe depression, severe anxiety or other psychiatric disorder referred to or undergoing special treatment, as judged by the investigator.
13. Severe sleep apnea (defined clinically).
14. Chronic diseases, as judged by the investigator.
15. Metformin treatment within 3 months prior to screening or concomitant medication influencing blood glucose (e.g. metformin and acarbose), influencing other parameters of metabolic syndrome (e.g. orlistat) or interfering with the investigational medicinal product.
16. Steroid treatment (oral or injected).
17. Concomitant medication addressing attention disorders.
18. Antidepressants that can lead to weight gain, as judged by the investigator.
19. Hypersensitivity to exenatide or to any of the excipients.
20. Pacemaker or metal implant that may interfere with Magnetic Resonance Imaging (MRI).
21. Claustrophobia (Uppsala and Salzburg) or abdominal diameter exceeding an MR gantry diameter of 70 cm (Salzburg).
22. Current or prior (within 3 months) participation in another clinical study involving an Investigational Medicinal Product (IMP).
23. A personal or family history of Medullary Thyroid Carcinoma (MTC)
24. A personal or family history of Multiple Endocrine Neoplasia syndrome type 2 (MEN 2).

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
BMI SDS (Body Mass Index Standard Deviation Score) | 6 months
  The primary objective is to compare the change from baseline to the 6 months visit, between lifestyle intervention + exenatide 2 mg once weekly and lifestyle intervention + placebo, in BMI SDS (according to WHO) for adolescents with obesity.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Forslund, Assoc Prof, Principal Investigator — Uppsala University Hospital
Locations (2):
- Department of Pediatrics, Salzburg State Hospital, Paracelsus Medical University, Salzburg, Austria
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Stenlid R, Cerenius SY, Wen Q, Aydin BK, Manell H, Chowdhury A, Kristinsson H, Ciba I, Gjessing ES, Morwald K, Gomahr J, Heu V, Weghuber D, Forslund A, Bergsten P. Adolescents with obesity treated with exenatide maintain endogenous GLP-1, reduce DPP-4, and improve glycemic control. Front Endocrinol (Lausanne). 2023 Nov 1;14:1293093. doi: 10.3389/fendo.2023.1293093. eCollection 2023. PMID 38027106